CLINICAL TRIAL: NCT02172378
Title: Effect of a 12-week Treatment With Inhaled Tiotropium (18 mcg Once Daily) on Lung Function and Static Lung Volumes in Stable, Moderate to Severe COPD Patients. Correlation to Dyspnoea Scales. A Double-blind, Placebo-controlled, Randomized, Parallel Group Study
Brief Title: 12-week Treatment With Inhaled Tiotropium (18 mcg Once Daily) on Lung Function and Static Lung Volumes in Stable, Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD) Patients. Correlation to Dyspnoea Scales
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.215
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (2):
- Tiotropium inhalation capsules (Experimental)
  Interventions: Drug: Tiotropium inhalation capsules
- Placebo inhalation capsules (Placebo Comparator)
  Interventions: Drug: Placebo inhalation capsules

INTERVENTIONS:
Drug: Tiotropium inhalation capsules
  Arms: Tiotropium inhalation capsules
Drug: Placebo inhalation capsules
  Arms: Placebo inhalation capsules

SUMMARY:
Determine the effect of 12-week treatment with inhaled tiotropium bromide on lung function and static lung volumes, correlate this effect with dyspnoea in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 40 years of age or older.
2. All patients had to have a diagnosis of COPD and had to meet the following spirometric and static lung volume criteria:

   1. Patients had to have relatively stable, moderate to severe airway obstruction with:

      * FEV1 ≤ 50 % of predicted value,
      * FEV1/SVC ≤ 70 %.
   2. All patients had to have the presence of lung hyperinflation as demonstrated by RV ≥ 125 % of predicted value.

   Predicted normal values were calculated according to European Community Coal and Steel (ECCS)

   Males:
   * FEV1 predicted (L) = 4.30 x height (metres) - 0.029 x age (years) - 2.49
   * RV predicted (L) = 1.31 x height (metres) + 0.022 x age (years) - 1.23

   Females:
   * FEV1 predicted (L) = 3.95 x height (metres) - 0.025 x age (years) - 2.60
   * RV predicted (L) = 1.81 x height (metres) - 0.016 x age (years) - 2.00
3. Patients had to be current or ex-smokers with a smoking history of more than 10 pack-years (p.y.). Patients who never smoked cigarettes were excluded.

   Number of p.y. = Number of cigarettes/day / 20 x years of smoking
4. Patients had to be able to perform all study related tests including the SWT, acceptable pulmonary function tests including PEFR measurements, and had to be able to maintain records during the study period as required in the protocol.
5. Patients had to be able to inhale medication from the HandiHaler.
6. All patients had to sign an informed consent form prior to participation in the trial i.e. prior to pre-study washout of their usual pulmonary medication.
7. Eosinophilia < 600/mm³ documented in the past year (if not available, a blood count cell was performed).

Exclusion Criteria:

1. Patients with a history of asthma, allergic rhinitis or atopy.
2. Patients with significant diseases other than COPD were excluded. A significant disease was defined as a disease which in the opinion of the investigator may have either put the patient at risk because of participation in the study or a disease which may have influenced the results of the study or the patient's ability to participate in the study.
3. Patients with a recent history (i.e. one year or less) of myocardial infarction.
4. Patients with a recent history (i.e. three years or less) of heart failure, pulmonary oedema, or patients with cardiac arrhythmia requiring drug therapy.
5. Patients who regularly used daytime oxygen therapy for more than one hour per day and in the investigator.s opinion was unable to abstain from the use of oxygen therapy.
6. Patients with known active tuberculosis.
7. Patients with a history of cancer within the last five years. Patients with treated basal cell carcinoma were allowed.
8. Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis.
9. Patients who underwent thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reason were evaluated as per exclusion criterion No. 2.
10. Patients with lower respiratory tract infection in the past six weeks prior to the Screening Visit (Visit 1) or during the run-in period.
11. Patients who were currently in a pulmonary rehabilitation programme or who completed a pulmonary rehabilitation programme in the six weeks prior to the Screening Visit (Visit 1).
12. Patients with known hypersensitivity to anticholinergic drugs, lactose or any other components of the inhalation capsule delivery system.
13. Patients with known symptomatic prostatic hypertrophy or bladder neck obstruction.
14. Patients with known narrow-angle glaucoma.
15. Patients who were treated with β-blockers, cromolyn sodium or nedocromil.
16. Patients who were treated with antihistamines (H1 receptor antagonists) or antileukotrienes.
17. Patients who were treated with monoamine oxidase inhibitors or tricyclic antidepressants.
18. Patients using oral corticosteroid medication at unstable doses (i.e. less than six weeks on a stable dose) or at a dose in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day.
19. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (i.e. oral contraceptives, intra-uterine devices, diaphragm or subdermal implants).
20. Patients with history and/or active significant alcohol or drug abuse.
21. Patients who took another investigational drug within one month or ten half lives (whichever was greater) prior to Visit 1.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2000-05; Primary Completion 2002-01 (Actual)

PRIMARY OUTCOMES:
trough FVC response at the end of the 12-week study | after 12 weeks of treatment (day 84)

SECONDARY OUTCOMES:
Determination of breathlessness (dyspnoea) as measured by the modified Borg scale | Screening, day 0, day 42, day 84
Evaluation of the Expiratory Flow Limitation (EFL) using the Negative Expiratory Pressure (NEP) method (optional) | Screening, day 0, day 42, day 84
Evaluation of inspiratory capacity (IC) | Screening, day 0, day 42, day 84, day 98
Evaluation of slow vital capacity (SVC) | Screening, day 0, day 42, day 84, day 98
Evaluation of FEV1 (Forced expiratory volume in one second) | Screening, day 0, day 42, day 84, day 98
Evaluation of FVC (Forced vital capacity) | Screening, day 0, day 42, day 84, day 98
Evaluation of FEF25-75% (Forced Expiratory Flow, mid expiratory phase) | Screening, day 0, day 42, day 84, day 98
Evaluation of FEF50% (Forced Expiratory Flow, at 50% of FVC) | Screening, day 0, day 42, day 84, day 98
Evaluation of FEF75% (Forced Expiratory Flow, at 75% of FVC) | Screening, day 0, day 42, day 84, day 98
Evaluation of thoracic gas volume (TGV) | Screening, day 0, day 42, day 84, day 98
Evaluation of dyspnoea by Baseline Dyspnoea index (BDI)/Transition Dyspnoea index (TDI) | Day 0, day 42, day 84
Evaluation of physician's global assessment | Day 0 (60 min. before dosing), day 42, day 84
Evaluation of COPD symptom scores (wheezing, shortness of breath, coughing and tightness of chest) | Day 0 (60 min before dosing), day 42, day 84
Amount of salbutamol therapy used during the trial period | 16 week evaluation period
Peak expiratory flow rate (PEFR) measured by the patients at home twice daily | 16 week evaluation period
Evaluation of Saint George's hospital respiratory questionnaire (SGRQ) | Day 0 (60 min. before dosing), day 42, day 84
Evaluation of Shuttle Walking test (SWT) | Screening, Day 0, day 42, 84
Occurence of adverse events | up to 14 weeks after treatment
Change from baseline in pulse rate (PR) in conjunction with spirometry at clinic visits | 16 weeks evaluation period
Change from baseline in blood pressure (BP) in conjunction with spirometry at clinic visits | 16 week evaluation period
Evaluation of total lung capacity (TLC) | Screening, day 0, day 42, day 84, day 98
Evaluation of flow resistance in the airways (Raw) | Screening, day 0, day 42, day 84, day 98
Evaluation of conductance of the airways (SGaw) | Screening, day 0, day 42, day 84, day 98
Evaluation of residual volume (RV) | Screening, day 0, day 42, day 84, day 98